CLINICAL TRIAL: NCT06369467
Title: A Phase 1 Dose-Escalation Study in Adults With Severe IgE-Mediated Food Allergy, to Assess the Safety, Tolerability, and Pharmacodynamic Effects of Short-Term Linvoseltamab Treatment, a BCMAxCD3 Bispecific Antibody to Induce T-Cell Killing of IgE Producing Plasma Cells, on Top of Chronic Dupilumab Treatment, to Prevent the Formation of New IgE Producing Plasma Cells
Brief Title: Short-Term Linvoseltamab Treatment on Top of Chronic Dupilumab Treatment for Adults With Severe Immunoglobulin E (IgE)-Mediated Food Allergy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5458-668-ALG-2219; 2024-511032-27-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Food Allergy
Keywords: Severe Immunoglobulin E (IgE)-Mediated Food Allergy; Peanut; Hazelnut; Walnut; Cashew; Milk; Egg/egg white; Soy; Wheat; Sesame; Cod; Salmon; Tuna; Lobster; Crab; Shrimp
MeSH Terms: conditions — Food Hypersensitivity; SeSAME syndrome | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Severe IgE-mediated food allergy (Experimental)
  Interventions: Drug: linvoseltamab; Drug: dupilumab

INTERVENTIONS:
Drug: linvoseltamab — Administered by intravenous (IV) infusion
  Other Names: REGN5458
Drug: dupilumab — Administered by subcutaneous (SC) injection
  Other Names: Dupixent®; REGN668

SUMMARY:
This study is researching an experimental drug called linvoseltamab combined with another drug called dupilumab. The study is looking at patients who have severe IgE-mediated food allergy. If the patient has an allergy, the body's defense system (immune system) overreacts to an allergen (eg, certain foods like peanuts, milk, shellfish) by making antibodies called IgE. An antibody is a protein that allows the immune system to find and fight off things the body does not recognize (allergens). IgE antibodies are sent out by cells like plasma cells. These antibodies and allergens bind to other cells that send out chemicals, causing an allergic reaction. The aim of the study is to see what side effects happen when linvoseltamab is combined with dupilumab.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drugs
* Does linvoseltamab combined with dupilumab affect other types of antibodies in the blood at different times
* How much study drug(s) is in the blood at different times

ELIGIBILITY:
Key Inclusion Criteria:

1. Clinical history of documented, ongoing, severe IgE-mediated allergy to food (peanut, hazelnut, walnut, cashew, milk, egg/egg white, soy, wheat, sesame, cod, salmon, tuna, lobster, crab and/or shrimp; documented symptom[s] of anaphylaxis due to exposure)
2. History of physician reported anaphylaxis to food requiring epinephrine administration and/or requiring an emergency visit or inpatient hospitalization
3. Participants with dupilumab-indicated atopic dermatitis (AD) must be receiving DUPIXENT as standard of care for the treatment of AD for a minimum of 12 weeks prior to screening OR Participants with dupilumab-indicated eosinophilic esophagitis (EoE) must be receiving DUPIXENT as standard of care for the treatment of EoE for a minimum of 12 weeks prior to screening OR Must be willing to initiate dupilumab treatment for food allergy
4. Participants initiating dupilumab treatment must agree to remain on dupilumab for the duration of the combination study treatment and safety follow-up periods. Participants who elect to enter the linvoseltamab re-dosing period, must also remain on continuous dupilumab treatment as outlined. Participants on commercial DUPIXENT must agree to remain on their prescribed dose, as described in the protocol, for the duration of the combination study treatment period
5. Participant must be willing to use an epinephrine auto-injector device
6. Participant must be willing to receive booster and/or re-vaccination(s), including for live (attenuated) vaccinations, based on results of vaccine antibody titers and investigator opinion
7. Has a body mass index between 18 and 32 kilogram per square metre (kg/m2), inclusive

Key Exclusion Criteria:

1. Pregnant or breastfeeding women
2. History of chronic disease (other than AD or EoE) requiring therapy (eg, heart disease, diabetes, hypertension) that, in the opinion of the principal investigator, would represent a risk to the participant's health or safety in this study or the participant's ability to comply with the study protocol. Participants on DUPIXENT for conditions other than AD or EoE (eg, asthma, chronic rhinosinusitis with nasal polyps, prurigo nodularis, etc) are excluded
3. Known or suspected progressive multifocal leukoencephalopathy (PML), or history of PML, neurodegenerative condition, central nervous system (CNS) movement disorder, or seizure within 12 months prior to Day 1
4. Recent history (within past 30 days) of a grade 3 or grade 4 gastrointestinal bleed, history of inflammatory bowel disease or severe diverticulitis or previous gastrointestinal perforation
5. History of moderate or severe asthma based on the Global Initiative for Asthma (GINA) guidelines
6. Pre-bronchodilator forced expiratory volume in the first second (FEV1) <80% of predicted using local reference values
7. Any prior exposure to a B-cell maturation antigen (BCMA) targeted therapy
8. Use of systemic corticosteroids within 2 months prior to screening
9. Use of other forms of allergen immunotherapy (eg, oral, SC, patch, or sublingual) or immunomodulatory therapy (not including corticosteroids) within 4 months prior to screening
10. Unwilling to discontinue use of antihistamines within 5 days prior to screening and within 5 days prior to skin prick test (SPT)
11. Hypersensitivity to epinephrine and any of the excipients in the epinephrine product
12. Within the previous 2 months of the screening visit has a history of bacterial, protozoal, viral or parasite infection requiring hospitalization or treatment with IV anti-infectives
13. Known history of human immunodeficiency virus (HIV) infection or HIV seropositivity at the screening visit

NOTE: Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2028-03-28 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From the initial first dose of linvoseltamab through the end of week 30
Severity of TEAEs | From the initial first dose of linvoseltamab through the end of week 30
Incidence of Adverse Event of Special Interest (AESIs) | From the initial first dose of linvoseltamab through the end of week 30
Severity of AESIs | From the initial first dose of linvoseltamab through the end of week 30
Incidence of Serious Adverse Events (SAEs) | From the initial first dose of linvoseltamab through the end of week 30
Severity of SAEs | From the initial first dose of linvoseltamab through the end of week 30

SECONDARY OUTCOMES:
Absolute change in the serum concentration of total IgE over time | Baseline to the end of week 30
Percent change in the serum concentration of total IgE over time | Baseline to the end of week 30
Time to reach unquantifiable total serum IgE concentration | Through the end of week 30
Time to reach baseline level and/or the lower limit of the normal ranges of serum IgG | Through the end of week 30
Time to reach baseline level and/or the lower limit of the normal ranges of serum immunoglobulin M (IgM) | Through the end of week 30
Time to reach baseline level and/or the lower limit of the normal ranges of serum immunoglobulin A (IgA) | Through the end of week 30
Incidence of participants with unquantifiable concentrations of serum total IgE | Through the end of week 30
Absolute change in the serum concentration of food allergen-specific IgE | Baseline through the end of week 30
  In participants who tested positive for a measured food allergen-specific IgE at baseline
Percent change in the serum concentration of food allergen-specific IgE | Baseline through the end of week 30
  In participants who tested positive for a measured food allergen-specific IgE at baseline
Time to reach unquantifiable food allergen-specific serum IgE levels | Through the end of week 30
  In participants who tested positive for a measured food allergen-specific IgE at baseline
Incidence of TEAEs | Following the combination study treatment period up to approximately 176 weeks
Severity of TEAEs | Following the combination study treatment period up to approximately 176 weeks
Incidence of AESIs | Following the combination study treatment period up to approximately 176 weeks
Severity of AESIs | Following the combination study treatment period up to approximately 176 weeks
Incidence of SAEs | Following the combination study treatment period up to approximately 176 weeks
Severity of SAEs | Following the combination study treatment period up to approximately 176 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (7):
- United States (5):
  - University of South Florida, Tampa, Florida
  - Emory University- Winship Cancer Institute, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Spain (2):
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Clinica Universidad de Navarra- Pamplona, Pamplona

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/